CLINICAL TRIAL: NCT06915376
Title: Comparison of Noninvasive Continuous Blood Pressure Measurement Using Artificial Intelligence-Assisted Pulse Oximetry and Electrocardiography Signal Combination With Invasive Arterial Blood Pressure
Brief Title: "AI-Based Noninvasive Blood Pressure Monitoring Compared to Invasive Arterial Measurement"
Acronym: NICONPRESS-1
Status: Completed | Type: Observational
Sponsor: Nevsehir Public Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif Yazar, MD, Associate Professor, Konya City Hospital
Other Study IDs: TABED-1-25-1137
Record Dates: First submitted 2025-03-28; First posted 2025-04-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Blood Pressure Measurement
Keywords: Noninvasive Blood Pressure Monitoring; Photoplethysmography; Artificial Intelligence; Intraoperative Hemodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Observational Cohort: This study includes a single group of adult patients undergoing elective non-cardiac surgery under general anesthesia. All participants will receive standard invasive arterial blood pressure monitoring. Simultaneously, noninvasive blood pressure data will be collected using the CPES (Combined Pulse Oximeter and ECG Signals) system. The study aims to compare the accuracy of CPES measurements to invasive values within the same individuals. No randomization or assignment to separate intervention groups will occur.
  Interventions: Device: CPES Monitoring

INTERVENTIONS:
Device: CPES Monitoring — Noninvasive blood pressure data will be collected using a combined pulse oximeter and ECG signal system (CPES) during elective non-cardiac surgery under general anesthesia. This system is used for observational purposes and does not alter the standard of care. The goal is to compare CPES-derived blood pressure values with invasive arterial blood pressure measurements.

SUMMARY:
The goal of this clinical trial is to evaluate a new, noninvasive method for continuously measuring blood pressure during surgery. This method combines two common types of signals - pulse oximetry and electrocardiography (ECG) - and uses artificial intelligence (AI) to help improve accuracy. Researchers will compare this method to the standard invasive arterial blood pressure (IABP) monitoring to see if it can safely and effectively replace invasive measurements in certain situations.

In surgeries, keeping blood pressure stable is extremely important. Sudden drops (hypotension) or spikes (hypertension) in blood pressure can cause serious organ problems after surgery. That's why continuous blood pressure monitoring is necessary, especially during key moments like anesthesia induction, intubation, and surgical positioning. In high-risk patients, clinicians often use invasive monitoring by inserting a catheter into an artery. While accurate, this method can cause complications, including bleeding, infection, blood clots, and in rare cases, damage to the limb. Studies show that blood clots can occur in nearly 20% of radial arterial lines, and up to 15% of cases experience bleeding or hematoma. Even life-threatening problems such as limb ischemia and embolism still occur in about 1% of patients.

Because of these risks, noninvasive continuous blood pressure measurement (NCBPM) devices are needed. Pulse oximeters, which are already used in all surgeries, measure oxygen in the blood and produce a waveform called photoplethysmography (PPG). This waveform changes with each heartbeat and reflects blood volume and flow. It can provide useful cardiovascular information, and in recent years, researchers have explored using PPG to estimate blood pressure. However, PPG alone may not give accurate results in all patients or conditions.

One reason for this is that important heart-related signals - like the time between heartbeats (R-R interval), the heart's pumping strength, and electrical conduction - are not captured by PPG alone. These signals are available through ECG. By combining ECG with PPG, researchers hope to get a more complete understanding of each heartbeat, and use this to estimate blood pressure more accurately.

In this study, the new combined method is called CPES (combined pulse oximeter and ECG signals). It uses signals from both devices, analyzed by artificial intelligence, to generate continuous blood pressure readings. The study will compare these readings with direct invasive arterial blood pressure values.

The main question the study aims to answer is:

Can CPES accurately measure systolic and diastolic blood pressure within 5 mmHg of the invasive method? This threshold is based on international standards (AAMI) for acceptable accuracy in blood pressure monitoring during surgery.

Secondary questions include:

Can CPES track rapid blood pressure changes during critical moments, such as after anesthesia drugs are given, during laryngoscopy, intubation, and surgical maintenance? Does the accuracy of KPES stay the same when the surgical table is tilted 15 degrees up (reverse Trendelenburg) or down (Trendelenburg)? These positions are commonly used in surgery and may affect blood pressure measurements.

Participants in this study will be adult patients undergoing general anesthesia. All participants will:

Have standard invasive arterial monitoring during surgery Wear ECG electrodes and a pulse oximeter Be monitored in real time using both standard and experimental systems Be placed in different surgical positions (as tolerated) for short periods to evaluate effects on blood pressure measurement Data will be collected at various stages of surgery and in different positions. The study does not change routine care but adds additional, noninvasive sensors for research purposes.

This study may help develop safer and more comfortable ways to measure blood pressure continuously during surgery. If successful, this method could reduce the need for invasive lines in many patients, lowering the risk of complications and making surgery monitoring easier and more cost-effective. It may also be useful in settings where invasive monitoring is not possible, such as emergency departments or outpatient procedures.

DETAILED DESCRIPTION:
Intraoperative blood pressure management plays a critical role in preventing postoperative complications, including organ dysfunction. While oscillometric intermittent noninvasive techniques are the standard for blood pressure monitoring in most surgical patients, they may fail to capture rapid hemodynamic fluctuations, especially during high-risk periods such as induction, intubation, and sudden positioning changes. In these cases, continuous invasive arterial blood pressure (IABP) monitoring is often used for real-time hemodynamic surveillance. However, IABP monitoring carries risks, including bleeding, thrombosis, hematoma, arterial occlusion, and bloodstream infections. Reported radial artery thrombosis rates reach as high as 19.7%, and catheter-related complications such as hematoma or bleeding occur in up to 15% of cases.

There is an increasing demand for noninvasive continuous blood pressure monitoring (NCBPM) technologies to avoid such complications. Photoplethysmography (PPG), derived from pulse oximeters, has emerged as a promising noninvasive technique. PPG waveforms reflect peripheral perfusion changes and offer insights into cardiac cycle dynamics. However, standalone PPG-based estimation is limited by its dependency on peripheral vascular tone, motion artifacts, and lack of electrical cardiac data.

To overcome these limitations, this study proposes a hybrid approach using synchronized photoplethysmography (PPG) and electrocardiography (ECG) signals, enhanced with artificial intelligence (AI)-based waveform analysis. This combination aims to improve the accuracy and temporal resolution of noninvasive continuous blood pressure monitoring. The proposed method, termed CPES (Combined Pulse Oximeter and ECG Signals), is based on the hypothesis that integrating electrical (ECG) and optical (PPG) signals will allow better modeling of arterial pulse wave velocity (PWV), pulse transit time (PTT), and surrogate hemodynamic parameters.

The study design includes intraoperative real-time recording of PPG and ECG signals in patients undergoing elective surgery under general anesthesia with concurrent IABP monitoring via radial artery catheterization. PPG waveforms will be acquired using a standard red/infrared dual-wavelength pulse oximeter (660 nm and 940-960 nm), and ECG will be collected using 3-lead continuous monitoring. Synchronization will be ensured using a time-stamping algorithm. Data acquisition will occur during distinct intraoperative phases: baseline (pre-induction), induction, intubation, maintenance, and positional interventions (±15° Trendelenburg and reverse Trendelenburg).

The primary outcome is the agreement between CPES-derived systolic and diastolic blood pressure values and simultaneously recorded invasive blood pressure values, assessed via Bland-Altman analysis. Clinical accuracy will be determined by comparing mean absolute error (MAE) and root mean square error (RMSE) to the AAMI/ANSI/ISO 81060-2 standard, which requires a mean difference of ≤5 mmHg and standard deviation of ≤8 mmHg.

Secondary outcomes include:

Ability of the CPES system to track rapid blood pressure changes (ΔSBP, ΔDBP) during induction and airway manipulation.

Evaluation of positional effects on blood pressure estimation accuracy using paired positional comparisons.

Exploratory modeling of derived hemodynamic parameters (e.g., PTT, HRV, PWV) and their correlations with arterial wave morphology and invasive BP metrics.

Signal processing will involve artifact removal, beat detection, normalization, and segmentation. Feature extraction will include time-domain, frequency-domain, and morphological features from both PPG and ECG. Machine learning models (e.g., gradient boosting, LSTM, or convolutional neural networks) may be trained on the dataset to enhance predictive performance.

This study aims to demonstrate that combining electrical and optical signals can yield clinically acceptable blood pressure measurements noninvasively, improving patient safety and reducing the need for invasive lines. If validated, this approach could be integrated into existing operating room monitors, expanding access to continuous BP monitoring in routine and resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for arterial catheter placement
* Age ≥18 years
* American Society of Anesthesiologists (ASA) physical status classification ≤3
* Planned surgical duration >60 minutes
* Non-cardiac surgery
* Expected supine positioning during the procedure
* Initial postoperative recovery planned in the Post-Anesthesia Care Unit (PACU)

Exclusion Criteria:

* Refusal to give informed consent
* Severe peripheral vascular disease
* Surgeries involving manipulation of major arteries
* Positive Allen's test
* Inability to place an arterial catheter in the upper extremity
* Presence of an arteriovenous fistula for hemodialysis
* Inability to measure NIBP (noninvasive blood pressure) on the same arm as the arterial catheter
* Difference greater than 10 mmHg in SBP or DBP between the two arms based on NIBP measurements
* Abnormal arterial pressure waveforms detected in history or initial IABP monitoring (e.g., pulsus paradoxus, pulsus alternans, pulsus bisferiens, pulsus parvus et tardus)
* Atrial fibrillation
* Body Mass Index (BMI) >35 kg/m²
* Preoperative hemoglobin level <10 g/dL or >16 g/dL
* Esophageal or nasopharyngeal pathology, or aortic coarctation
* Conditions affecting accurate pulse oximeter readings, such as nail or finger disorders (e.g., nail fungus or scleroderma), or presence of nail polish, dye, henna, or tattoos on fingers or nails.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from adult patients undergoing elective non-cardiac surgery under general anesthesia at Konya City Hospital. All participants will have a clinical indication for arterial catheter placement as part of routine intraoperative monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Primary Outcome-1: Accuracy of Noninvasive Systolic Blood Pressure Estimation Compared to Invasive Reference | Intraoperative period (from induction to surgical maintenance)
  The predicted systolic blood pressure values obtained from the combined pulse oximeter and ECG signal (CPES) system will be compared to invasive arterial blood pressure (IABP) measurements. Accuracy will be evaluated using the following statistical metrics:
  Mean Squared Error (MSE)
  Mean Absolute Error (MAE)
  Correlation Coefficient (R)
  Coefficient of Determination (R²)
2. Primary Outcome-2: Accuracy of Noninvasive Diastolic Blood Pressure Estimation Compared to Invasive Reference | Intraoperative period
  The predicted diastolic blood pressure values obtained from the CPES system will be compared to invasive arterial blood pressure (IABP) measurements. Accuracy will be assessed using:
  Mean Squared Error (MSE)
  Mean Absolute Error (MAE)
  Correlation Coefficient (R)
  Coefficient of Determination (R²)

SECONDARY OUTCOMES:
Secondary Outcome-1: Detection of Rapid Hemodynamic Changes During Critical Intraoperative Events | From anesthesia induction to 10 minutes after intubation
  This outcome will evaluate whether the CPES (Combined Pulse Oximeter and ECG Signals) system can detect rapid changes in blood pressure during key intraoperative phases, such as anesthesia induction, laryngoscopy, intubation, and early maintenance.
  The continuous blood pressure values estimated by CPES will be compared to real-time invasive arterial blood pressure (IABP) values recorded simultaneously.
  The system's ability to track hemodynamic fluctuations will be assessed by comparing the magnitude and timing of changes (ΔSBP and ΔDBP) between the two methods.
Secondary Outcome-2: Effect of Patient Position on Noninvasive Blood Pressure Estimation Accuracy | During intraoperative positional changes (Trendelenburg and reverse Trendelenburg)
  This outcome will assess whether patient positioning affects the accuracy of blood pressure readings obtained by CPES. Participants will be placed in 15-degree Trendelenburg and reverse Trendelenburg positions for 10 minutes each, as tolerated. At each position, systolic and diastolic blood pressure values estimated by CPES will be compared to invasive arterial blood pressure (IABP) readings.
  The goal is to determine whether CPES measurements change appropriately in response to gravitational and physiological changes due to body positioning, and whether they remain consistent with invasive reference measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Akif Yazar, MD, Principal Investigator — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Konya/Meram, Turkey (Türkiye)